CLINICAL TRIAL: NCT00875836
Title: Buspirone Treatment for Marijuana Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Aimee McRae-Clark, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01DA026782 (NIH); R01DA026782 (NIH); DPMCDA
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-07

CONDITIONS: Marijuana Dependence
Keywords: Marijuana; Buspirone; Contingency management; Motivational enhancement therapy
MeSH Terms: conditions — Marijuana Abuse | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buspirone (Experimental): Buspirone
  Interventions: Drug: Buspirone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buspirone — Flexible dose, up to 60 mg daily
  Other Names: Buspar
  Arms: Buspirone
Drug: Placebo — Flexible dose, up to 60 mg daily
  Arms: Placebo

SUMMARY:
Marijuana is the most commonly used illicit drug, yet few clinical trials have evaluated pharmacotherapy treatments for marijuana dependence. This study will evaluate the efficacy of buspirone for reducing marijuana use in marijuana-dependent adults. A contingency management (CM) intervention and motivational enhancement therapy (MET) will be incorporated to encourage study engagement and retention. It is hypothesized that buspirone combined with MET and CM will reduce the percent of marijuana-positive urine drug screen results in marijuana-dependent individuals as compared to a placebo treatment combined with MET and CM.

ELIGIBILITY:
Inclusion Criteria:

* Must meet DSM-IV criteria for marijuana dependence.
* Must be between the ages of 18 and 65 years.
* If female and of childbearing potential, must agree to use acceptable methods of birth control for the duration of the trial.
* Must consent to random assignment, and be willing to commit to psychosocial behavioral and medication treatment.
* Must be able to read and provide informed consent.

Exclusion Criteria:

* Women who are pregnant, nursing, or plan to become pregnant during the course of the study.
* Must not have a history of or current psychotic disorder, bipolar disorder, or eating disorder.
* Must not pose a current suicidal or homicidal risk.
* Must not meet current criteria for major depression.
* Must not have evidence or history of serious hematologic, endocrine, cardiovascular, pulmonary, renal, gastrointestinal or neurologic disease.
* Must not require concomitant therapy with psychotropic medication.
* Must not be currently dependent on other substances, with the exception of nicotine or caffeine.
* Hypersensitivity to buspirone or any other product component.
* Patients who, in the investigator's opinion, would be unable to comply with study procedures or assessments, or would be unacceptable study candidates (e.g., poses threat to staff).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2009-09; Primary Completion 2014-06 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee McRae-Clark, Pharm.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited between November 2009 and March 2014 primarily through media and internet advertisements.
Groups:
- Buspirone: Buspirone: Flexible dose up to 60 mg/day
- Placebo: Placebo: Flexible dose up to 60mg/day
Period: Overall Study
Arm/Group | Buspirone | Placebo
Started | 88 | 87
Completed | 45 | 47
Not Completed | 43 | 40

BASELINE CHARACTERISTICS:
Groups:
- Buspirone: Buspirone: 30 mg capsules twice daily
- Placebo: Placebo: 30 mg capsules twice daily
- Total: Total of all reporting groups
Arm/Group | Buspirone | Placebo | Total
Number analyzed (Participants) | 88 | 87 | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 88 | 87 | 175
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 67 | 67 | 134
Region of Enrollment [Number; unit: participants]
  United States | 88 | 87 | 175

OUTCOME MEASURES:

1. Primary Outcome: Percent Marijuana-negative Urine Drug Screens (UDS)
Description: Participants submitted a urine sample weekly. Percentage of marijuana negative urine samples were calculated per group.
Time Frame: Participants provided a once-weekly urine sample for twelve weeks
Measure: Number; unit: percentage of UDS
Units Other Than Participants: UDS samples
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 88 | 87
Number analyzed (UDS samples) | 1056 | 1044
percentage of UDS | 7.2 | 6.4

2. Secondary Outcome: Retention in the Study
Description: Number of days subjects remained active in the study
Time Frame: participants were followed for twelve weeks
Measure: Median (Inter-Quartile Range); unit: Day
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 88 | 87
Day | 79 [18 to 91] | 84 [14 to 91]

3. Secondary Outcome: Marijuana Craving
Description: The Marijuana Craving Questionnaire (MCQ) is intended to measure marijuana craving in adults. It measures symptoms on four subscales: expectancy, purposefulness, emotionality, and compulsivity. The scale rates individual items from 1 (least craving) - 7 (most craving) with a composite scoring range of 12-84 and possible subscale scoring range of 3-21. It was administered weekly- reported here is the mean composite score across the 8 week treatment course.
Time Frame: 8 Weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 88 | 87
units on a scale | 29.6 [27.0 to 32.2] | 28.4 [25.8 to 31.1]

ADVERSE EVENTS:
Arm/Group | Buspirone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/87
Other Adverse Events (participants affected / at risk) | 73/88 | 66/87
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buspirone (N=88) | Placebo (N=87)
Anxiety or Depression (Psychiatric disorders) | 4 (5) | 5 (5)
Dizziness or lightheaded (Nervous system disorders) | 36 (44) | 11 (17)
Drowsiness (Nervous system disorders) | 17 (19) | 15 (18)
Gastrointestinal (Gastrointestinal disorders) | 36 (61) | 23 (35)
Headache (Nervous system disorders) | 28 (55) | 27 (46)
Insomnia (Nervous system disorders) | 16 (17) | 15 (17)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 11 (19) | 24 (32)
Sinus/allergies/flu (General disorders) | 13 (19) | 12 (16)
Congestion (Respiratory, thoracic and mediastinal disorders) | 19 (26) | 18 (23)
Other (General disorders) | 43 (87) | 40 (83)

LIMITATIONS AND CAVEATS:
Limitations included significant attrition during the course of the 12-week trial, difficulty with UCT interpretation due to the long excretion half-life of marijuana in urine, and likelihood that the genetic analysis was underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No